CLINICAL TRIAL: NCT01649999
Title: Phase 2b Study of ASP015K - A Double-Blind, Placebo-Controlled, Dose-Finding Study in Moderate to Severe Rheumatoid Arthritis Patients
Brief Title: A Study to Evaluate the Efficacy and Safety of ASP015K in Moderate to Severe Rheumatoid Arthritis Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 015K-CL-RAJ1
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; ASP015K
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- ASP015K lowest dose (Experimental): Oral
  Interventions: Drug: peficitinib
- ASP015K low dose (Experimental): Oral
  Interventions: Drug: peficitinib
- ASP015K medium dose (Experimental): Oral
  Interventions: Drug: peficitinib
- ASP015K high dose (Experimental): Oral
  Interventions: Drug: peficitinib
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: peficitinib — oral
  Other Names: ASP015K
  Arms: ASP015K high dose; ASP015K low dose; ASP015K lowest dose; ASP015K medium dose
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy and safety of ASP015K monotherapy and to evaluate the dose-dependent response of ASP015K in moderate to severe Rheumatoid Arthritis (RA) subjects given ASP015K for 12 weeks.

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, double-blind, parallel-group, placebo-controlled, dose-finding, monotherapy, multi-center study with once daily oral ASP015K or matching placebo in subjects with moderate to severe RA, with or without prior antirheumatic medication, and regardless of responsiveness to the medication.

The study is comprised of up to a 4-week Screening period, a 12-week Treatment period and a 4-week Follow-up period.

Subjects in each treatment group will take ASP015K or matching placebo orally, once daily, after breakfast for 12 weeks after the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has received a full explanation of the study drug and this study in advance, and written informed consent to participate in the study has been obtained from the subject himself/herself
* Outpatient has RA that was diagnosed according to the 1987 revised criteria of the ACR at least 6 months prior to screening
* At screening subject has active RA as evidenced by all of the following:

  * ≥ 6 tender/painful joints;
  * ≥ 6 swollen joints;
  * CRP of ≥ 0.5 mg/dL or ESR of ≥ 28 mm/h.C-Reactive Protein (CRP) of ≥ 0.8 mg/dL or Erythrocyte Sedimentation Rate (ESR) of ≥ 28 mm/hr
* Subject meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA, Class I, II or, III at screening

Exclusion Criteria:

* Positive tuberculin (TB) test within 90 days of Screening
* Abnormal chest x-ray indicative of an acute or chronic infectious process or malignancy
* Receipt of live or live attenuated virus vaccination within 30 days prior to the first dose of study drug
* Hepatitis B virus or hepatitis C virus carrier or has a history of a positive test for human immunodeficiency virus (HIV) infection
* Any other autoimmune rheumatic disease, other than Sjogren's syndrome
* Previous history of clinically significant infections or illness (requiring hospitalization or requiring parenteral therapy) within 90 days of the Screening visit, or a history of any illness that would preclude participation in the study
* History of any malignancy, except for successfully treated basal or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix
* Does not meet specified washout criteria for the following RA medications: etanercept, certolizumab, adalimumab, golimumab, infliximab and tocilizumab, rituximab, abatacept, anakinra, methotrexate, sulfasalazine, hydroxychloroquine, gold, penicillamine or leflunomide
* Previous intolerance to Janus kinase (JAK) inhibitors
* Receipt of intra-articular or parenteral corticosteroid within 28 days prior to the first dose of study drug
* Receipt of plasma exchange therapy within 60 days prior to the start of study drug
* Receipt of any investigational agent within 30 days or 5 half-lives, whichever is longer, prior to first dose of study drug
* Receipt of medications that are CYP3A substrates with narrow therapeutic range within 14 days prior to first dose of study drug
* History of heart failure, defined as New York Heart Association (NYHA) grade 3 or greater

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2013-07-20 (Actual); Study Completion 2013-07-20 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving American College of Rheumatology Criteria 20 (ACR 20) response | Week 12

SECONDARY OUTCOMES:
Percentage of Subjects achieving ACR 50 response | Week 12
Percentage of Subjects achieving ACR 70 response | Week 12
Change from baseline in Disease Activity Score using 28 joint count and C Reactive Protein (DAS28-CRP) | Baseline and Week 12
Safety assessed by the incidence of adverse events, vital signs, 12-lead ECGs and clinical labo-tests | During 12-week treatment period and 4-week follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Tōhoku

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Toyoshima J, Kaibara A, Shibata M, Kaneko Y, Izutsu H, Nishimura T. Exposure-response modeling of peficitinib efficacy in patients with rheumatoid arthritis. Pharmacol Res Perspect. 2021 May;9(3):e00744. doi: 10.1002/prp2.744. PMID 33929089
- [Derived] Takeuchi T, Tanaka Y, Iwasaki M, Ishikura H, Saeki S, Kaneko Y. Efficacy and safety of the oral Janus kinase inhibitor peficitinib (ASP015K) monotherapy in patients with moderate to severe rheumatoid arthritis in Japan: a 12-week, randomised, double-blind, placebo-controlled phase IIb study. Ann Rheum Dis. 2016 Jun;75(6):1057-64. doi: 10.1136/annrheumdis-2015-208279. Epub 2015 Dec 15. PMID 26672064
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=334